CLINICAL TRIAL: NCT00832234
Title: Phase II Study of Combination Bortezomib, Dexamethasone, and Rituximab in Previously Untreated Patients With Waldenstroms Macroglobulinemia: A Multicenter Trial of the European Myeloma Network
Brief Title: Bortezomib, Dexamethasone, and Rituximab in Untreated Waldenstroms Macroglobulinemia
Acronym: BDR-WM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Myeloma Network B.V. (Network)
Collaborators: University of Athens (Other); University of Roma La Sapienza (Other); Niguarda Hospital (Other); University of Turin, Italy (Other); University of Salamanca (Other); Hospital Clinic of Barcelona (Other); Hotel Dieu Hospital (Other); Erasmus Medical Center (Other); University Hospital, Toulouse (Other); Fondazione IRCCS Policlinico San Matteo di Pavia (Other); Laikο General Hospital, Athens (Other); Klinikum der Universitaet Muenchen, Grosshadern (Other); Aalborg University Hospital (Other); Centre Hospitalier de Lens (Other); Universitaire Ziekenhuizen KU Leuven (Other); Theagenio Cancer Hospital (Other Government); University of Wuerzburg (Other); Skane University Hospital (Other); Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Professor Hans Erik Johnsen, Sponsor Office Director, Professor, European Myeloma Network B.V.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMN-01 (26866138CAN 2021); EudraCT-nr. 2006-003563-31
Record Dates: First submitted 2009-01-27; First posted 2009-01-30 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Waldenstroms Macroglobulinemia
Keywords: Morbus Waldenstrom; Waldenstroms Macroglobulinemia; Therapy; Rituximab; Dexamethasone; Bortezomib
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — Bortezomib; Dexamethasone; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BDR (Experimental)
  Interventions: Drug: Bortezomib, Dexamethasone, Rituximab

INTERVENTIONS:
Drug: Bortezomib, Dexamethasone, Rituximab — The combination of bortezomib, dexamethasone and rituximab will be administered in five treatment cycles. Bortezomib will be administered as an iv push over 3 to 5 seconds at a dose of 1.3mg/m2/day on days 1,4,8 and 11 of cycle one. On cycles 2-5 bortezomib will be given at a dose of 1.6mg/m2/day on days 1,8,15 and 22 of each cycle. Only on cycles 2 and 5, following the administration of bortezomib, dexamethasone 40mg IV and rituximab 375mg/m2 IV will be administered. A total of 8 infusions of rituximab will be administered. The administration of bortezomib before rituximab may abrogate the IgM flare phenomenon that occurs frequently after the first course of rituximab.
  Other Names: Velcade; MabThera

SUMMARY:
This is a Phase II multicenter study designed to evaluate the safety and efficacy of combination BDR. BDR will be administered in one 21-day treatment cycle followed by four 35-day treatment cycles to patients with WM.

DETAILED DESCRIPTION:
Title: Phase II Study of Combination Bortezomib (VELCADE, PS-341), Dexamethasone, and Rituximab (MabThera) (BDR) in Patients with previously untreated Waldenstroms Macroglobulinemia (WM).

Objectives:

The primary objective of this study is:

* To determine the response rate [the combined complete response (CR) + partial response (PR) + minimal response (MR)] following treatment with BDR in patients with previously untreated WM.

Secondary objectives are:

* To determine time to progression following treatment with BDR.
* To assess the safety and tolerability of BDR in patients with WM.

Patient population:

Patients with previously untreated WM who have an indication for treatment are candidates for the study.

Specific inclusion and exclusion criteria are detailed in the protocol.

Number of patients:

Sixty-one patients are to be enrolled in this multicenter study. This study will be conducted within centers participating in the European Myeloma Network.

Study design and methodology This is a Phase II multicenter study designed to evaluate the safety and efficacy of combination BDR. BDR will be administered in one 21-day treatment cycle followed by four 35-day treatment cycles to patients with WM. Bortezomib will be administered as an iv push over 3 to 5 seconds at a dose of 1.3mg/m2/day on days 1,4,8 and 11 of cycle 1. On cycles 2-5 bortezomib will be given at a dose of 1.6mg/m2/day on days 1,8,15 and 22 of each cycle. Only on cycles 2 and 5, following the administration of Bortezomib, dexamethasone 40mg iv and Rituximab 375 mg/m2 iv will be administered. A total of 8 infusions of rituximab will be administered. Subsequently patients rated as CR, PR, MR or SD will be followed without any treatment until there is evidence of progressive disease.

A Screening visit will be conducted within 28 days before baseline (baseline being Day 1, Cycle 1, before study drug administration). At this visit, a medical history will be obtained and a complete physical examination will be performed including vital signs, height, weight, and a 12-lead electrocardiogram. A neurological questionnaire will also be completed. Disease assessments will be performed, including performance status, bone marrow aspirate and biopsy, Beta2-microglobulin, serum protein electrophoresis with quantification of immunoglobulins and immunofixation studies, CT scanning of the chest, abdomen and pelvis. Clinical laboratory tests including a complete blood count plus differential, electrolytes, urea, creatinine, total bilirubin, SGOT (ALT), SGPT (AST), LDH, total protein and albumin. Patients who meet the eligibility requirements as assessed at the Screening visit will be enrolled in the study and start study drug treatment. Patients will be evaluated after each cycle with serum protein electrophoresis to determine their response to therapy. If patients demonstrate a response or have stable disease at the end of each cycle they will continue to receive therapy. If the patient demonstrates evidence of progressive disease at the end of each cycle then the patient will be removed from study. Modified response criteria updated at the Third International Workshop on Waldenstroms macroglobulinemia will be used to assess response, stable disease (SD), and progressive disease (PD) in this study. Changes of serum monoclonal protein concentration will be assessed from serum protein electrophoresis rather than from nephelometric measurement of serum immunoglobulins. Patients will receive five cycles of therapy. Subsequently, it is strongly advised that blood stem cells will be collected from patients <70 years of age for future high-dose therapy.

At the end of each cycle patients will have testing performed to assess for toxicity and efficacy. A directed questionnaire for neurologic toxicities, review of concomitant medications and other support therapies, including growth factors and transfusions will also be performed. Three months after the last dose of study drug, and every three months thereafter for 2 years, patients are to attend follow-up study visits. At these visits, a physical examination will be performed and Karnofsky performance status assessed. Patients will have a neurological questionnaire completed, have tests for disease assessments including serum and protein electrophoresis with quantification of immunoglobulins and immunofixation studies, Beta2-microglobulin, bone marrow aspirate and biopsy (only if the patient is in a complete remission), CT scanning of the chest, abdomen and pelvis (only if patient had evidence of WM disease on baseline scans). Serum and protein electrophoresis with quantification of immunoglobulins and immunofixation studies must be repeated > 6 weeks if a patient attains a complete response. At the follow-up study visits, a complete blood count plus differential, electrolytes, urea, creatinine, total bilirubin, SGOT, will also be obtained.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following inclusion criteria to be enrolled in this study:

* Clinicopathological diagnosis of Waldenstroms macroglobulinemia as defined by consensus panel one of the Second International Workshop on Waldenstroms macroglobulinemia.
* All patients with the diagnosis of WM will be evaluable for response according to the response criteria
* No prior systemic treatment for WM. Prior plasmapheresis to control hyperviscosity, is allowed. In that case baseline monoclonal protein levels for assessment of response will be the levels prior to plasmapheresis, if this is the higher value prior to treatment initiation
* Patients must have at least one of the following indications to initiate treatment as defined by Consensus Panel Two recommendations from the Second -
* International Workshop on Waldenstroms Macroglobulinemia.
* Recurrent fever, night sweats, weight loss, fatigue
* Hyperviscosity
* Lymphadenopathy which is either symptomatic or bulky (>5cm in maximum diameter)
* Symptomatic hepatomegaly and/or splenomegaly
* Symptomatic organomegaly and/or organ or tissue infiltration
* Peripheral neuropathy due to WM
* Symptomatic cryoglobulinemia
* Cold agglutinin anemia
* Immune hemolytic anemia and/or thrombocytopenia
* Nephropathy related to WM
* Amyloidosis related to WM
* Hemoglobin < 10g/dL
* Platelet count < 100x109/L
* Serum monoclonal protein >5g/dL even with no symptoms
* CD20 positive disease based on any previous bone marrow immunohistochemistry or flow cytometric analysis performed up to 3 months prior to enrollment.
* Karnofsky performance status more than 60.
* Life-expectancy >3 months.
* Baseline platelet count more than 50x109/L, and absolute neutrophil count more than 0.75x109/L.
* Meet the following pretreatment laboratory criteria at the Screening visit conducted within 28 days of study enrollment:

  * AST (SGOT): less than 3 times the upper limit of institutional laboratory normal.
  * ALT (SGPT): less than 3 times the upper limit of institutional laboratory normal.
* Total Bilirubin: less than 2 times the upper limit of institutional laboratory normal, unless clearly related to the disease.
* Calculated or measured creatinine clearance: less than 30 mL/minute. Serum sodium >130 mmol/L.
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion Criteria:

* Patients meeting any of the following exclusion criteria are not to be enrolled in the study.
* Prior systemic treatment with WM (plasmapheresis is allowed)
* Myocardial infarction within 6 months prior to enrollment or has New York
* Hospital Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Patient has hypersensitivity to dexamethasone, bortezomib, boron or mannitol.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Cardiac amyloidosis
* Peripheral neuropathy or neuropathic pain grade 2 or higher as defined by NCI - CTCAE version 3
* Women who are pregnant.
* Women who are breast-feeding and do not consent to discontinue breast-feeding.
* Women of childbearing age who are not willing to use effective anti-conceptive methods for the duration of the study and 6 months thereafter.
* Men who do not consent not to father a child during the treatment period and six months thereafter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2006-09; Primary Completion 2010-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The response rate [the combined complete response (CR) + partial response (PR) + minimal response (MR)] following treatment with BDR in patients with previously untreated WM. | Two years

SECONDARY OUTCOMES:
Time to progression following treatment with BDR The safety and tolerability of BDR in patients with WM. | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Meletios A Dimopoulos, MD, Principal Investigator — University of Athens School of Medicine, Alexandra Hospital, Athens, Greece
Locations (1):
- University of Athens School of Medicine, Athens, Greece